CLINICAL TRIAL: NCT01846468
Title: A Partially-blinded, Randomized, Placebo-controlled, Adaptive Single and Multiple Ascending Dose Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of LHW090 in Healthy Volunteers and in Subjects With Renal Dysfunction
Brief Title: An Ascending Dose Study to Assess Safety, Tolerability, PK/PD of LHW090 in Healthy Volunteers and in Subjects With Renal Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CLHW090X2101
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2017-02

CONDITIONS: Chronic Renal Insufficiency
Keywords: Healthy volunteers and patients,; renal insufficiency,
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Stage 1 : LHW090, Healthy Volunteers (Experimental): Healthy Volunteers will receive single dose of LHW090 on Day 1.
  Interventions: Drug: LHW090
- Stage 2: LHW090, Healthy Volunteer (Experimental): Healthy Volunteers across 7 single ascending dose cohorts will be administered LHW090 or matching placebo day 1
  Interventions: Drug: LHW090; Drug: Placebo
- Stage 3: LHW090, Healthy Volunteer (Experimental): Healthy Volunteers across 6 multiple ascending dose cohorts will be administered LHW090 or matching placebo for 14 days.
  Interventions: Drug: LHW090; Drug: Placebo
- Stage 4: LHW090, Patients (Experimental): Subjects with Chronic Renal Insufficiency across 3 cohorts will be administered a single dose of LHW090 in Day 1.
  Interventions: Drug: LHW090

INTERVENTIONS:
Drug: LHW090 — 1 mg, 12.5 mg, 100 mg capsules
Drug: Placebo — Matching placebo capsules
  Arms: Stage 2: LHW090, Healthy Volunteer; Stage 3: LHW090, Healthy Volunteer

SUMMARY:
The purpose of the study is to provide pertinent information to enable decisions regarding the developability of LHW090 for use in patients with chronic renal insufficiency, including a comparison of the potential risk-benefit ratio of several doses of the study drug to enable optimal doses to be tested in later studies.

ELIGIBILITY:
Inclusion Criteria: For Stage 1, 2 and 3 subjects only:

Subjects eligible for inclusion in these stages of the study have to fulfill all of the following criteria at screening:

* Healthy male and female subjects age 18 to 45 years of age included, and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
* At screening, and first baseline, vital signs (systolic and diastolic blood pressure and pulse rate) will be assessed in the sitting position after the subject has rested for at least three minutes, and again (when required) after three minutes in the standing position. Sitting vital signs should be within the following ranges:

oral body temperature between 35.0-37.5 °C systolic blood pressure, 90-140 mm Hg diastolic blood pressure, 50-90 mm Hg pulse rate, 40 - 90 bpm

For Stage 4 subjects only:

* Male and female subjects, age 18 to 75 years of age included, with previously identified chronic renal insufficiency (estimated or measured GFR ≤ 45ml/min/1.73m2, or diabetic with estimated or measured GFR ≤ 60ml/min/1.73m2.) Diabetes can be established by the prescription and current use of anti-glycemic drugs, a random fasting glucose level of ≥ 144mg/dl or a hemoglobin A1c of ≥ 6.5%
* At screening, vital signs (systolic and diastolic blood pressure and pulse rate) will be assessed in the sitting position after the subject has rested for at least three minutes, and again (when required) after three minutes in the standing position. Sitting vital signs should be within the following ranges:

oral body temperature between 35.0-37.5 °C systolic blood pressure, 90-179 mm Hg diastolic blood pressure, 50-100 mm Hg pulse rate, 40 - 95 bpm

Exclusion Criteria:

For Stages 1, 2 and 3, subjects fulfilling any of the following additional criteria are not eligible for inclusion in this study:

* An active history of clinically significant ECG abnormalities as determined by the Investigator, or any of the following ECG abnormalities at Screening or Baseline:
* Long QT syndrome
* QTcF > 450 msec (males; at screening)
* QTcF > 460 msec (females; at screening)
* Known history of current clinically significant arrhythmias.
* Use of phosphodiesterase-5 inhibitors, UNLESS subjects agree to discontinue use of the drug for the duration of the study.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant
* Smokers (use of tobacco products in the previous 3 months). Urine cotinine levels will be measured during screening and at each baseline for all subjects. Smokers will be defined as any subject who reports tobacco use and/or who has a urine cotinine ≥ 500 ng/ml.
* Hemoglobin levels below 11.0 g/dl at screening.
* Subjects in Stage 3 only of the study will be excluded if they have any of the following:
* A history of allergy to topical anesthetic drops
* A history of corneal disease
* A history of eye surgery within three months prior to screening
* A history of corneal surgery (including refractive surgery and corneal transplantation)

For Stage 4, subjects fulfilling any of the following additional criteria are not eligible for inclusion in this study:

* An active history of clinically significant ECG abnormalities as determined by the Investigator, or any of the following ECG abnormalities at Screening or Baseline:
* Long QT syndrome
* QTcF > 480 msec at screening
* Use of phosphodiesterase-5 inhibitors, UNLESS subjects agree to discontinue use of the drug for the duration of the study.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant
* Significant smokers. Significant smokers who are unable to tolerate using no more than 4 cigarettes a day should be excluded
* History of right ventricular dysfunction within the last 12 months
* Hemoglobin levels below 9.0 g/dl at screening.
* Use of angiotensin converting enzyme inhibitors (ACEi), UNLESS subjects agree to either a withholding of their ACEi, or a switch to an angiotension receptor blocker, starting 5 days (or 5 half-lives which ever is longer) prior to initiation of study and extending to the end-of-study visit. Patient who withhold their ACEi for the specified duration must first consult with their primary physician to determine their suitability and safety for this temporary withholding of ACEi.
* Diuretic-dependence, i.e. unable to produce urine without diuretics, or at high risk of flash pulmonary edema without diuretics. Use of diuretics will exclude subjects UNLESS subjects agree to withhold diuretics starting the day prior to check-in and extending to discharge. Consultation of the subject with their primary physician must be used to determine their suitability and safety for temporary withholding of their diuretics.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2014-06-28 (Actual); Study Completion 2014-06-28 (Actual)

PRIMARY OUTCOMES:
Number of participants (Healthy Volunteers) with reported adverse events receiving single oral dose of LHW090 as assessment of safety and tolerabiility | 6 months
  In this analysis AE and SAE will be reported
Number of participants (Healthy Volunteers) with reported adverse events receiving multiple oral dose of LHW090 as assessment of safety and tolerabiility | 6 months
  In this analysis AE and SAE will be reported
Number of participants (patients) with reported adverse events receiving single oral dose of LHW090 as assessment of safety and tolerabiility | 6 months
  In this analysis AE and SAE will be reported

SECONDARY OUTCOMES:
Pharmacokinetics of LHW090/LHV527 in plasma: observe maximum plasma concentration following LHW090 at steady state in healthy volunteers and patients | Within 60 min prior to dosing, post dose: +/- 5 min up to 3 hrs, +/- 10 min from ≥3 hrs to 24hrs, +/- 2 hrs from ≥24 hrs to 72hrs
  In this analysis Cmax will be reported
Pharmacokinetics of LHW090/LHV527 in plasma: time to reach the maximum concentration after administration of LHW090 (Tmax) | Within 60 min prior to dosing, post dose: +/- 5 min up to 3 hrs, +/- 10 min from ≥3 hrs to 24hrs, +/- 2 hrs from ≥24 hrs to 72hrs
  In this analysis Tmax will be reported
Pharmacokinetics of LHW090/LHV527 in plasma: area under the plasma concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) | Within 60 min prior to dosing, post dose: +/- 5 min up to 3 hrs, +/- 10 min from ≥3 hrs to 24hrs, +/- 2 hrs from ≥24 hrs to 72hrs
  In this analysis AUClast will be reported
Pharmacokinetics of LHW090/LHV527 in plasma: area under the plasma concentration-time curve from time zero to infinity (AUCinf) | Within 60 min prior to dosing, post dose: +/- 5 min up to 3 hrs, +/- 10 min from ≥3 hrs to 24hrs, +/- 2 hrs from ≥24 hrs to 72hrs
  In this analysis AUCinf will be reported
Pharmacokinetics of LHW090/LHV527 in plasma: terminal elimination half-life (T1/2) | Within 60 min prior to dosing, post dose: +/- 5 min up to 3 hrs, +/- 10 min from ≥3 hrs to 24hrs, +/- 2 hrs from ≥24 hrs to 72hrs
  In this analysis T1/2 will be reported
Pharmacokinetics of LHW090/LHV527 in plasma: accumulation ratio (RACC) | Within 60 min prior to dosing, post dose: +/- 5 min up to 3 hrs, +/- 10 min from ≥3 hrs to 24hrs, +/- 2 hrs from ≥24 hrs to 72hrs
  In this analysis the accumulation ratio will be reported
Pharmacokinetics of LHW090/LHV527 in plasma: apparent volume of distribution during the terminal elimination phase following extravascular administration (Vd/F) | Within 60 min prior to dosing, post dose: +/- 5 min up to 3 hrs, +/- 10 min from ≥3 hrs to 24hrs, +/- 2 hrs from ≥24 hrs to 72hrs
  In this analysis apparent volume of distribution during the terminal elimination phase will be reported
Pharmacokinetics of LHW090/LHV527 in plasma: apparent system clearance from plasma following intravenous administration of iothalamate (CL/F) | Within 60 min prior to dosing, post dose: +/- 5 min up to 3 hrs, +/- 10 min from ≥3 hrs to 24hrs, +/- 2 hrs from ≥24 hrs to 72hrs
  In this analysis the apparent system clearance from plasma will be reported
Pharmacokinetics of LHW090/LHV527 in urine: apparent system clearance from urine from time 0 - 24 hrs following drug administration (Ae0-24) | Stage 1, 2 and 4 :0-4, 4-8, 8-12, 12-24, 24-36, 36-48 and 48 - 72 h post dose in Day 1 and Day 14; Stage 3: 0-4, 4-8, 8-12, and 12-24 h post dose
  In this analysis the apparent system clearance by urine will be reported from 0 - 24 hrs post dose
Pharmacokinetics of LHW090/LHV527 in urine: apparent system clearance from urine from time 0 - 72 hrs following drug administration (Ae0-72h) | Stage 1, 2 and 4 :0-4, 4-8, 8-12, 12-24, 24-36, 36-48 and 48 - 72 h post dose in Day 1 and Day 14; Stage 3: 0-4, 4-8, 8-12, and 12-24 h post dose
  In this analysis the apparent system clearance by urine will be reported from 0 - 72 hrs post dose
Pharmacokinetics of LHW090/LHV527 in urine: apparent renal clearance from urine following drug administration (CLr) | Stage 1, 2 and 4 :0-4, 4-8, 8-12, 12-24, 24-36, 36-48 and 48 - 72 h post dose in Day 1 and Day 14; Stage 3: 0-4, 4-8, 8-12, and 12-24 h post dose
  In this analysis the apparent system clearance by urine will be reported
Pharmacodynamics of LHW090/LHV527 in serum: post treatment peak and mean area under the plasma concentration-time curve from time zero to 24 hour (AUC0-24h/24h) for cyclic guanosine (cGMP) | Within 60 min prior to dosing, post dose: +/- 5 min up to 3 hrs, +/- 10 min from ≥3 hrs to 24hrs, +/- 2 hrs from ≥24 hrs to 72hrs
  In this analysis AUC0-24/24h will be reported for single ascending dose healthy volunteers and CRI subjects
Pharmacodynamics of LHW090/LHV527 in serum: post treatment peak and mean area under the plasma concentration-time curve from time zero to 24 hour (AUC0-24h/24h) for atrial natriuretic peptide (ANP) | Within 60 min prior to dosing, post dose: +/- 5 min up to 3 hrs, +/- 10 min from ≥3 hrs to 24hrs, +/- 2 hrs from ≥24 hrs to 72hrs
  In this analysis AUC0-24/24h will be reported for single ascending dose healthy volunteers and CRI subjects

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- United States (2):
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Knoxville, Tennessee

REFERENCES:
- See also: Results for CCLHW090X2101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=15009